CLINICAL TRIAL: NCT03688750
Title: Impact of Different Shoe Heel Heights on Spinal Configuration During Different Phases of Menstrual Cycle
Brief Title: Impact of Different Shoe Heel Heights on Spinal Configuration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, HAhmed, lecturer of biomechanics, Cairo University
Other Study IDs: P.T.REC/012/001884
Record Dates: First submitted 2018-09-02; First posted 2018-09-28 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2018-11

CONDITIONS: Impact of Different Heel Heights on Spinal Configuration
Keywords: heel height; spinal configuration; phases of menstrual cycle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention

SUMMARY:
90 healthy female subjects with regular menstrual cycle ,their ages ranged from 19-25 years,their BMI ranged from 18-25 will be participated in this study.

Formetric Raster Stereography will be used to assess spinal configuration while each participant wear shoes of different heel heights 2.5 cm (low),4.5 cm (moderate) and 7 cm (height) during early follicular and mid luteal phases of menstrual cycle.

DETAILED DESCRIPTION:
* this study will be conducted on healthy females to investigate effect of different heel heights footwear on spine posture and pelvic position by using formetric 4 D analysis system which is a light-optical scanning method based on Video-Raster-Stereography (VRS). Accordingly, the system consists of a light projector which projects a line grid on the back of the patient which is recorded by an imaging unit. A computer software analyzes the line curvature that generates from it. the formetric provides comprehensive information about the whole body statics and posture in only one measuring process, e.g. spine curvature (lateral and frontal), vertebral rotation, and pelvic position.
* There is generally no need for reflecting markers, because the anatomical fixed points Vertebra prominens (VP), Sacrum Point (SP), Dimple Left (DL) Dimple Right (DR) as well as the spinal center line and spinal rotation are automatically detected by the system. That allows a very time-saving and reliable examination procedure.
* shoe characteristics: standard shoes will be used and designed to fit females in sizes ranging from 37-41 and different heel heights (2.5 cm low, 4,5 cm moderate and 7 cm high).
* Descriptive statistics including mean and standard deviation will be applied for dependent variables and participant demographics. repeated measures analysis of variance will be implemented to detect the difference in dependent measures among three heel condition.

ELIGIBILITY:
Inclusion Criteria:

* Their ages ranged from 19-25.
* Their BMI ranged from 18-25
* They wear high heeled shoes occasionally for less than 10 H/week or not at all
* they are able to wear high heel without pain.

Exclusion Criteria:

* any female with spinal deviation,previous spinal surgeries,leg length discrepancy or foot deformities
* Joint stiffness, ankle sprain
* any case with orthopedic or neurological problems
* Females with irregular menstrual cycle

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 90 healthy females with regular menstrual cycle
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
kyphotic angle | from 9/2018 to 6/2019
  this the maximum angle measured between surface tangents of the upper inflection point in the vicinity of the vertebra prominence and the thoracic lumbar inflection point
Lordotic angle | from 9/2018 to 6/2019
  this the maximum angle measured between surface tangents of the thoracic lumbar inflection point and lower lumbar-sacral inflection point
trunk imbalance | from 9/2018 to 6/2019
  trunk imbalance is defined as the lateral deviation of the vertebra prominence from the mid line dimple
trunk inclination | from 9/2018 to 6/2019
  trunk inclination refers to a difference in the height between vertebra prominence and dimple mid line based on a vertical plane (sagittal section)
pelvic tilting | from 9/2018 to 6/2019
  pelvic tilt refers as the difference in the height of the lumbar dimple based on horizontal plane ( transverse section)
pelvic inclination | from 9/2018 to 6/2019
  it is calculated as the mean torsion of the dimple left and dimple right surface normals